CLINICAL TRIAL: NCT02690116
Title: Effects of Meditative Movement (Qigong/Tai Chi Easy) on Fatigued Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: University of Arizona (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1R01CA182901-01A1 (NIH)
Record Dates: First submitted 2016-01-06; First posted 2016-02-24 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Fatigue
Keywords: Meditative movement; Breast cancer survivors; Qigong; Tai Chi Easy; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Training Support

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Qigong/Tai Chi Easy (Experimental): The Qigong/Tai Chi Easy (QG/TCE) intervention has been standardized, manualized, and has a formal training program for instructors from the Institute of Integral Qigong and Tai Chi (IIQTC).
  Interventions: Other: Qigong/Tai Chi Easy
- Sham Qigong (Sham Comparator): This active control group uses a gentle movement intervention, with similar types of movements with the same energy expenditure, but without the meditative states and breath focus as QG/TCE (validated in the pilot study using the Meditative Movement Inventory).
  Interventions: Other: Sham Qigong
- Educational Support (Active Comparator): The Recovery Support Group will consist of a classroom-style intervention, designed to educate, engage interaction, and maintain participation and attention over 8 weeks. This group will include readings/discussions specific to breast cancer, and social interaction facilitation.
  Interventions: Other: Educational Support

INTERVENTIONS:
Other: Qigong/Tai Chi Easy — Classes will be at two different times of day (to accommodate working and non-working participants). Participants will attend one 60 minute class per week for the 8 weeks, with a recommended home practice time of 2 1/2 hours each week.
  Arms: Qigong/Tai Chi Easy
Other: Sham Qigong — Classes will be at two different times of day (to accommodate working and non-working participants). Participants will attend one 60 minute class per week for the 8 weeks, with a recommended home practice time of 2 1/2 hours each week.
  Arms: Sham Qigong
Other: Educational Support — Class times and at-home readings correspond to dose set for the QG/TCE and SQG class times and home practice. Participants will attend one 60-minute class per week for the 8 weeks, with a recommended home practice time (reading, workbook completion) of 2 1/2 hours each week.
  Arms: Educational Support

SUMMARY:
The purpose of this study is to test whether Meditative Movement (based on a standardized and tested Qigong/Tai Chi Easy protocol) is more efficacious for improving fatigue and other symptoms in women after treatment for breast cancer than (a) a non-meditative "sham" Qigong active intervention and (b) an inactive education / support group.

DETAILED DESCRIPTION:
Patients with breast cancer often report fatigue and other associated symptoms that persist for months, even years, after treatment ends. In a recent pilot study of Qigong/Tai Chi Easy (QG/TCE, a low-intensity form of Meditative Movement), fatigued breast cancer survivors experienced greater improvements in fatigue (medium effect size, .56); compared to a "sham" Qigong control intervention (also low-intensity activity). Trends for improvement compared to control were found for sleep quality and depression. Recruitment for the single-site implementation was steady, and feasible. To build upon the promise of this pilot study, and to further test intervention components that may elucidate what aspects of the intervention have the most impact, a three-group, randomized trial will be undertaken to test effects of an 8-week QG/TCE intervention on fatigue and other symptoms at the end of 8 weeks, and 24 weeks post-intervention. 246 (attrition to 210) women who are 6 months to 10 years past treatment for Stage 0- III breast cancer, aged 45-75, and post-menopausal, will be randomized into one of three study arms. Two comparison groups will be used, an educational support (ES) group control and an active sham Qigong (SQG) group with movements that are similar to and with the same level of physical activity intensity as QG/TCE, but without the focus on the breath and meditative state. These treatments allow for separation of effects associated with gentle exercise alone (controlled in SQG) and education/social support alone without any exercise (controlled in ES) relative to the mind-body practice of QG/TCE, to distinguish unique effects of the meditative and breath foci. The study will be implemented in two sites in a large, metropolitan area, including one low-income hospital (and catchment neighborhood) with larger numbers of Latina survivors where our research team has extensive community connections and cultural experience implementing exercise and meditative movement programs. Psychometrics and biomarkers related to symptoms before and after the interventions will be examined to further our understanding of the mechanisms associated with effects of QG/TCE, as distinct from ES and SQG.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer, stage 0-III
* Between 6 months and 10 years past primary treatment
* Post-menopausal
* Experiencing fatigue (scoring < 75 on "Vitality" scale of Short Form (SF)-36)
* English-speaking or Spanish-speaking

Exclusion Criteria:

* Women who are unable to stand for 10-minute segments
* Women who have had substantial experience with mind-body practices that blend movement with mindfulness/breathing techniques, such as Yoga, Tai Chi, or Qigong
* Women who work night shifts (fatigue-related factor)
* Restless leg syndrome (fatigue-related factor)
* Hypothyroidism (fatigue-related factor)
* Currently diagnosed with anemia (fatigue-related factor)
* Uncontrolled diabetes (fatigue-related factor)
* Major severe clinical depression (fatigue-related factor)
* Use of antihistamine, cyclosporins, corticosteroids, sleeping aids
* Regular use of alcohol (more than 2 drinks per day)

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Fatigue Symptom Inventory | Change from baseline fatigue to fatigue at 8 weeks and fatigue at 6 months.
  Fatigue

SECONDARY OUTCOMES:
Profile of Mood States Short Form (POMS-SF) | Change from baseline anxiety and depression to anxiety and depression at 8 weeks and anxiety and depression at 6 months.
  Anxiety and depression
Functional Assessment of Cancer Therapy-Cognitive Function (FACT-COG) | Change from baseline cognitive function to cognitive function at 8 weeks and cognitive function at 6 months.
  Cognitive function
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline sleep quality to sleep quality at 8 weeks and sleep quality at 6 months
  Sleep quality
Women's Health Initiative Brief Physical Activity Questionnaire (WHI-BPAQ) | Change from baseline physical activity (PA) to PA at 8 weeks and PA at 6 months
  Physical activity
Venipuncture for serum using MILLIPLEX MAP Human Cytokine/Chemokine Magnetic Bead Panel kits | Change from baseline Inflammatory biomarkers (IL-1β, IL-6,TNF-α; IFN-γ) to Inflammatory biomarkers at 8 weeks
  Inflammatory biomarkers (IL-1β, IL-6,TNF-α; IFN-γ)
Diurnal salivary samples (enzyme assay) | Change from baseline salivary cortisol to salivary cortisol at 8 weeks
  Salivary cortisol
ActiGraph GT3X activity monitor | Change from baseline objective physical activity to objective physical activity at 8 weeks and objective physical activity at 6 months
  Objective measurement of physical activity
ActiGraph GT3X activity monitor | Change from baseline objective sleep quality to objective sleep quality at 8 weeks and objective sleep quality at 6 months
  Objective measurement of sleep quality

OTHER OUTCOMES:
Functional Assessment of Cancer Therapy-Cognitive Function Neuropathy (FACT-COGNtx) | Change from baseline peripheral neuropathy to peripheral neuropathy at 8 weeks and peripheral neuropathy at 6 months
  Peripheral Neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Linda Larkey, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No